CLINICAL TRIAL: NCT05254483
Title: ACTIWEB-PA (Active Children Through In-home Web-based Physical Activity): a Feasibility Trial of a Youth Targeted, Web-based Physical Activity Intervention.
Brief Title: Web-based Physical Activity Intervention for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-0504; A176000 (Other: UW, Madison); EDUC/KINESIOLOGY/KINESIOLOG (Other: UW, Madison); Protocol ver 4.0 04-01-2021 (Other: UW, Madison)
Record Dates: First submitted 2022-02-23; First posted 2022-02-24 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Physical Activity in Children
Keywords: Web based physical activity tools; Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental): Receiving exercise program immediately
  Interventions: Behavioral: UNICEF kid power program immediately; Device: ActiGraph Accelerometer
- Waitlist Control Group (WCG) (Active Comparator): Receiving exercise program after 12 week wait.
  Interventions: Behavioral: UNICEF kid power program for waitlist control; Device: ActiGraph Accelerometer

INTERVENTIONS:
Behavioral: UNICEF kid power program immediately — The intervention will be delivered via the UNICEF Kid Power website (https://www.unicefkidpower.org/) and any screened device such as a computer, smartphone, smart TV or an electronic tablet can be used to watch the videos and perform the assigned physical activity.
  Participants will self-select activities 5 days a week. The participants will have the choice to undertake the physical activity in bouts and accumulate it over the course of the day.
  To promote adherence to intervention, a weekly email with reminder to perform the physical activity will be sent to parents. In addition, research-based articles on the importance of physical activity and behavior change in children will also be emailed.
  Arms: Intervention group (IG)
Behavioral: UNICEF kid power program for waitlist control — The wait-list control group will perform physical activity as usual and will only receive a weekly email on the importance of healthy dietary habits in children. The intervention will last 12 weeks. At the end of the study, the wait-list control group will be offered the UNICEF Kid Power intervention for a duration of 12-weeks
  Arms: Waitlist Control Group (WCG)
Device: ActiGraph Accelerometer — The participants will be mailed accelerometers and instructed to wear for 7 consecutive days during their waking hours, prior to the start of intervention. The mail containing the accelerometer will accompany pictorial instructions, explaining in detail the correct way of wearing it.

SUMMARY:
The purpose of this study is to conduct a two-arm randomized controlled trial and evaluate the feasibility, acceptability, and effects on the physical and psychosocial outcomes of children in response to a web-based physical activity intervention. 80 participants aged 8-11 will be enrolled in the Madison, WI area and can expect to be on study for up to 12 weeks.

DETAILED DESCRIPTION:
The COVID-19 pandemic has facilitated the broadening of the landscape of the physical activity (PA) programs offered to children. This has been due to the fact that, traditional school-based PA offerings and other organized sport programs were on a nearly a year long hiatus. In the absence of structured PA, web-based PA programs for children garnered approval from families because of the safety and convenience offered. It is anticipated that the web-based exercise programs will remain appealing even after the pandemic is over, and may coexist with the in-person PA offerings. These programs will likely persist due to the convenience offered, the increasing penetration of 'smart' screen-based devices, and increasing usage of internet in American homes. The examples of web-based PA programs for children include, educational websites based on behavior change theories, mobile-app based PA programs, and web-based exercise videos. Of these, the latest to enter the web-based PA space and the most under-researched are the exercise videos based programs. Web-based, exercise videos feature a 'follow-after-me' format encouraging children to enact the movements shown. Examples of a few popular programs offering such videos are UNICEF Kid Power, GoNoodle, and CosmicKids Yoga.

There have been no formal evaluations of web-based, exercise video programs for children so far. Moreover, there have been very few evaluations of other types of web-based PA interventions. Even fewer evaluations have addressed the impact of such programs on children's quality of life and psychosocial health. Investigators will fill this research gap by conducting a pilot trial examining the feasibility of the previously untested, exercise video based, UNICEF Kid Power intervention. Study team will also determine the effects of the program on physical and psychosocial health outcomes. Doing so will help investigators to compute the sample size of the future full-scale trial, and to optimize it based on the learnings from the pilot trial.

Specific Aims

Aim 1 (Primary aim): To examine the feasibility of the processes involved in implementing the UNICEF Kid Power intervention by measuring recruitment, retention, and intervention adherence rates.

Aim 2: To examine the safety, acceptability, and satisfaction with the intervention using qualitative measures.

Aim 3: To determine effect sizes for outcomes of physical activity, physical function, psychosocial health, and self-concept to facilitate estimation of sample size for a future full-scale randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Insufficient physical activity (not meeting the federal physical activity guideline of 60 min/day of moderate-to-vigorous intensity physical activity or at least 3 days per week of muscle strengthening or at least 3 days per week of bone strengthening activities as part of the daily 60 min/day of PA)
* Availability of internet in the household
* Availability of a smart-phone/computer/electronic tablet in the household
* Ability of the participant and a parent to communicate in English language

Exclusion Criteria:

* Developmental (autism), learning (dyslexia) and mental health disorders (ADHD, oppositional defiant disorder, depression, anxiety, and other mental health disorders) as diagnosed by a physician
* Parent reported disability/impairments that would interfere with the child's ability to safely perform the exercises in the videos. These include motor and sensory disabilities and impairment.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Feasibility: Percentage of Participants Recruited | up to 12 weeks
  Proportion of recruited will be computed by dividing the number of participants recruited into the study by those who completed the screener and met the eligibility criteria. This proportion will then be converted into a percentage. A priori target of 50% recruitment rate will be set.
Retention Rate: Percentage of Participants Completing 12 week Intervention | up to 12 weeks
  Retention rate will be computed as the percentage of randomized participants completing 12-week assessments. A priori target of 80% retention rate will be set.
Adherence Rate: Percentage of Participants Performing Physical Activity (PA) on 70% of assigned Videos | up to 12 weeks
  Adherence to intervention will be monitored as a measure of implementation fidelity. This will be expressed as the percentage of participants performing PA on 70% of the assigned videos each week of the intervention period.

SECONDARY OUTCOMES:
Change in average number of steps per day | Baseline and 12 weeks (post intervention)
  Physical activity will be assessed by measuring average step counts per day by pedometer at baseline and 12-weeks. Parents will be reporting children's step-count in an online log at the end of every day.
Score on Physical functioning and psychosocial health questionnaire (PedsQL)- child reported | Baseline and 12 weeks (post intervention)
  PedsQL assesses four dimensions of health: physical functioning, social functioning, emotional functioning, and school functioning. The latter three dimensions can also be aggregated to create a "psychosocial health summary score." The scale is an ideal choice because it addresses a broad range of psychosocial domains including emotional aspects related to symptoms of anxiety and sadness. Because PedsQL scale is designed to be interviewer-administered, it will be completed by the children during a videocall with the study coordinator.
  It is a 23 item scale. Each item can be answered on a scale of "0-4" where 0 - never a problem, 1 - Almost never a problem, 2- Sometimes a problem, 3 - Often a problem, 4 - Almost always a problem. Higher scores indicate worse physical and psychological health.
Change in Score on Piers-Harris Children's Self-Concept Scale | Baseline and 12 weeks (post intervention)
  Piers-Harris Children's Self-Concept Scale (3rd ed) assesses self-concept and comprises 58 items and six domains. Children/adolescents indicate whether each item applies to them by selecting a yes or no response. Raw scores are converted to standardized T-scores. Higher scores indicate favorable self-concept whereas lower scores mean lower self-concept in both global and domain-specific scales.

OTHER OUTCOMES:
Change in Study Participation Experience Survey (Quantitative) | 6 weeks (mid intervention) and 12 weeks (post intervention)
  The investigators will conduct a short mid-study survey (at 6 weeks) which will be repeated at 12 weeks, and will be completed by a parent. This survey will assess feasibility of uptake of the intervention and the challenges encountered. The quantitative portion of the survey includes 6-items scored on a 4-point likert scale (for a range of 0-24 where higher scores indicate barriers to participation).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cadmus-Bertram, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No